CLINICAL TRIAL: NCT06597656
Title: An Open-Label, Systemic Gene Delivery Study to Evaluate the Safety, Tolerability and Expression of Delandistrogene Moxeparvovec Following Plasmapheresis in Subjects With Duchenne Muscular Dystrophy and Pre-existing Antibodies to AAVrh74
Brief Title: A Gene Transfer Therapy to Evaluate the Safety and Efficacy of Delandistrogene Moxeparvovec (SRP-9001) Following Therapeutic Plasma Exchange (Plasmapheresis) in Participants With Duchenne Muscular Dystrophy (DMD) and Pre-existing Antibodies to AAVrh74
Acronym: HORIZON
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study is being terminated due to a business decision.
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRP-9001-105
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Gene-Delivery; DMD; Ambulatory; Pediatric; Duchenne; Seropositive; Pre-existing antibodies; AAVrh74 antibody; Plasmapheresis; Titer; Seropositivity
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Delandistrogene Moxeparvovec After Plasmapheresis Procedure (Experimental): Participants will receive a single intravenous (IV) infusion of delandistrogene moxeparvovec on Day 1 after plasmapheresis procedure if AAVrh74 antibodies are sufficiently low.
  Interventions: Genetic: delandistrogene moxeparvovec; Procedure: Plasmapheresis

INTERVENTIONS:
Genetic: delandistrogene moxeparvovec — Single IV infusion of delandistrogene moxeparvovec
  Other Names: SRP-9001; delandistrogene moxeparvovec-rokl; ELEVIDYS
Procedure: Plasmapheresis — Therapeutic plasma exchange procedure

SUMMARY:
This is a gene transfer therapy study evaluating the safety of and delandistrogene moxeparvovec dystrophin protein expression from delandistrogene moxeparvovec following therapeutic plasma exchange (plasmapheresis) in ambulatory male participants with DMD and pre-existing antibodies to AAVrh74 over a period of 59 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory per protocol specified criteria.
* Has a definitive diagnosis of DMD prior to Screening based on documentation of clinical findings and prior confirmatory genetic testing.
* Ability to cooperate with motor assessment testing.
* Has elevated AAVrh74 antibody titers per protocol-specified requirements.
* A pathogenic frameshift mutation, nonsense mutation or premature stop codon or pathogenic variant in the DMD gene that is expected to lead to absence of dystrophin protein with exception of a mutation in exon 8 and/or 9.
* Stable daily dose of oral corticosteroids for at least 12 weeks prior to Screening, and the dose is expected to remain constant throughout the study (except for modifications to accommodate changes in weight).

Exclusion Criteria:

* Has reduced left ventricular ejection fraction on the screening ECHO or clinical signs and/or symptoms of cardiomyopathy.
* Presence of any other clinically significant illness, including cardiac, pulmonary, hepatic, renal, hematologic, immunologic, or behavioral disease, or infection or malignancy or concomitant illness or requirement for chronic drug treatment that in the opinion of the Investigator creates unnecessary risks for gene transfer or a medical condition or extenuating circumstance that, in the opinion of the Investigator, might compromise the participant's ability to comply with the protocol required testing or procedures or compromise the participant's wellbeing, safety, or clinical interpretability.
* Exposure to gene therapy, investigational medication, or other protocol-specified treatment within the protocol specified time limits.
* Abnormality in protocol-specified diagnostic evaluations or laboratory tests. .

Note: Other inclusion or exclusion criteria could apply.

Ages: 4 Years to 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Quantity of Delandistrogene Moxeparvovec Dystrophin Expression Adjusted by Muscle Content Biopsied Muscle as Measured by Western Blot | Baseline, Week 12
Change From Baseline in Quantity of Delandistrogene Moxeparvovec Dystrophin Expression in Biopsied Muscle as Measured by Immunofluorescence (IF) Fiber Intensity | Baseline, Week 12
Change From Baseline in Quantity of Delandistrogene Moxeparvovec Dystrophin Expression in Biopsied Muscle as Measured by IF Percent Dystrophin-positive Fibers (PDPF) | Baseline, Week 12
Mean Concentration of Vector Genome Copies Using Polymerase Chain Reaction in Muscle Tissue Biopsy, After Delandistrogene Moxeparvovec Administration | Week 12

SECONDARY OUTCOMES:
Number of Participants with a Treatment Emergent Adverse Event (TEAE), Adverse Event of Special Interest (AESI), and Serious Adverse Event (SAE) | Baseline up to End of Study (Up to Week 59)
Change from Baseline in rAAVrh74 Antibody Titers | Baseline, Week 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (3):
- United States (3):
  - University of Florida, College of Medicine, Gainesville, Florida
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio